CLINICAL TRIAL: NCT04303416
Title: Effect of Plasma Exchange With Albumin in Patients With Adrenomyeloneuropathy: Unicentric, Single Arm, Proof of Concept Study.
Brief Title: Plasma Exchange With Albumin in AMN Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pujol, Aurora, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XAMNPEAP2019
Record Dates: First submitted 2020-03-06; First posted 2020-03-11 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Adrenomyeloneuropathy; Adrenoleukodystrophy
Keywords: plasma exchange; albumin; VLCFA
MeSH Terms: conditions — Adrenoleukodystrophy | interventions — Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental): Patients before and after the treatment
  Interventions: Drug: Albumin solution

INTERVENTIONS:
Drug: Albumin solution — plasma exchange with albumin, one per week for one month, then one per month for 5 months
  Other Names: plasma exchange

SUMMARY:
Adrenoleukodystrophy (X-ALD) is the most common genetic disorder of the brain white matter with an incidence of 1:14,700 births. It is caused by mutations in the ABCD1 gene, which encodes a transporter of very long-chain fatty acids (VCLFA) into the peroxisome for degradation. As a consequence VLCFA accumulate in tissues and plasma being the pathognomonic biomarker for diagnosis. The excess of VLCFA produces mitochondrial ROS and oxidative damage, a major factor driving X-ALD pathogenesis. Other key dysregulated pathways are energy production, mitochondrial biogenesis and respiration, proteostasis, and ER stress. Current therapeutic options are unsatisfactory, restricted to bone marrow transplant and gene therapy, for which most patients do not qualify. The encouraging results of plasma exchange (PE) with albumin replacement for Alzheimer's Disease prompted us to start this study. Our rationale is the following: In plasma, VLCFA are transported by lipoproteins and albumin. Albumin is the major transporter of fatty acids (FA) to the brain. ABCD1 deficiency induces inflammation and increases blood-brain barrier leakage, which could facilitate increased permeability to albumin. We posit that replacement of albumin would lower VLCFA levels in plasma through peripheral sink mechanisms, diminishing the quantity of VLCFA reaching the brain, and would prevent lipid peroxidation. A pilot proof-of-concept study in 5 X-ALD patients will be carried out to replace endogenous albumin through PE applied, once a week the first month and monthly for 5 months. A 6 months follow-up after the end of the treatment will be carried out.

ELIGIBILITY:
Inclusion Criteria:

1. Men of 18 to 65 years old, inclusive
2. Elevated plasma VLCFA and gene mutation identified
3. Clinical signs of AMN with at least pyramidal signs in the lower limbs and difficulties to run
4. Presence of motor deficit according to the EDSS scale
5. Ability to perform the 2MWT
6. Normal brain MRI or brain MRI showing the following abnormalities that can be observed in AMN patients without the cerebral form of X-ALD, obtained in the 6 months prior to screening:

   * abnormal hyperintensity of pyramidal tract fibers in the brain stem on FLAIR or T2 sequence
   * abnormal hyperintensity of pyramidal tract fibers in the internal capsules on FLAIR or T2 sequence
   * cerebellar atrophy
   * moderate cortical atrophy

Exclusion Criteria:

1. Any contraindication for plasma exchange due to behavioral disorders or abnormal coagulation parameters, such for example:

   * Hypocalcemia (Ca++ < 8.7 mg/dl)
   * Thrombocytopenia (< 100.000/µl)
   * Fibrinogen < 1.5 g/l
   * Prothrombin time (Quick) p< 60% versus control (INR > 1.5)
   * Beta-blocker treatment and bradycardia < 55/min
   * Treatment with ACIs (increased risk of allergic reactions)
2. Hemoglobin < 10 g/dl
3. Difficult venous access precluding plasma exchange
4. A history of frequent adverse reactions (serious or otherwise) to blood products
5. Hipersensibility to albumin o allergies to any of the components of Albunorm® 5%
6. Plasma creatine > 2 mg/dl
7. Uncontrolled high blood pressure (systolic blood pressure of 160 mmHg or higher and/or diastolic blood pressure of 100 mmHg or higher despite regular treatment during the last 3 months)
8. Liver cirrhosis or any liver problem with GPT > 2.5 x ULN, or bilirubin > 2 mg/dl
9. Heart diseases as evidenced by myocardial infarction, severe or unstable angina, or heart failure in the past 12 months
10. Gadolinium enhancement on T1 sequence of any abnormal hypersignal of white matter, including myelinated pyramidal tracts, visible at brain MRI on FLAIR sequences
11. Significant peripheral edema (2+ or more on the Assessment Chart for Pitting Edema) of the extremities of any etiology
12. Any evolutive malignancy during the last five years or any condition complicating adherence to the study protocol
13. Smokers (one pack/ day or more for at least 20 years), current or former
14. Any psychiatric disease
15. Present participation to another therapeutic clinical trial for X-ALD, or the receipt of any other investigational drug in the three months prior to the start of the study
16. Patients being treated with anticoagulants or antiplatelet therapy
17. Not easily contactable by the investigator in case of emergency or not capable to call the investigator

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Concentration of very long chain fatty acids | Change from baseline at 6 months
  Concentration of C26:0, C24:0 fatty acids and C26:0/C22:0 ratio in plasma

SECONDARY OUTCOMES:
2 Minute Walk Test | Months 0, 6 and 12
  It measures the distance an individual is able to walk over a total of two minutes on a hard, flat surface
6 Minute Walk Test | Months 0, 6 and 12
  It measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface
Timed Up and Go (TUG) test | Months 0, 6 and 12
  It consists in standing up, walking 3 meters, turning around, walk back to the chair and sitting back down, at regular pace
Time to walk 25 Feet (TW25) | Months 0, 6 and 12
  The patient should walk 7.62 meters (25 feet) as quickly, but safely, as possible without running
Expanded disability status scale (EDSS) | Months 0, 6 and 12
  This scale measures motor function, ranging from 0 (normal neurological examination) to 10 (death)
Ashworth scale | Months 0, 6 and 12
  The Modified Ashworth Scale measures spasticity in patients with lesions of the CNS or neurological disorders. It ranges from 0 (no increase in tone) to 4 (affected part(s) rigid in flexion or extension).
SF-Qualiveen (Short-form Qualiveen) | Months 0, 6 and 12
  The Qualiveen is a specific patients' health-related quality of life developed to assess the impact of urinary disorders in patients with neurological conditions. Response options are framed as 5-point Likert-type scales, with 0 indicating no impact of urinary problems on health-related quality of life and 4 indicating a high adverse impact.

CONTACTS AND LOCATIONS:
Locations (1):
- Bellvitge University Hospital, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided